CLINICAL TRIAL: NCT00882024
Title: A Phase II, Randomized Multi-Center, Double-Blind Study of Tranilast With Concomitant Methotrexate (MTX) Compared to MTX Alone in Patients With Active Rheumatoid Arthritis (RA)
Brief Title: Safety and Efficacy Study of Tranilast in Patients With Active Rheumatoid Arthritis (RA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nuon Therapeutics, Inc. (Industry)
Responsible Party: Michael Kitt, MD/Chief Medical Officer, Nuon Therapeutics, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A3003RA
Record Dates: First submitted 2009-04-14; First posted 2009-04-16 (Estimated); Last update posted 2011-01-06 (Estimated); Status verified 2011-01

CONDITIONS: Active Rheumatoid Arthritis
Keywords: Rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tranilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 Tranilast (Experimental): Tranilast, 300 mg/day
  Interventions: Drug: Tranilast
- 2 Tranilast (Experimental): Tranilast, 150 mg/day
  Interventions: Drug: Tranilast
- 3 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranilast — 150 mg tranilast tablets, bid, 12 weeks
  Arms: 1 Tranilast
Drug: Tranilast — 75 mg tablets, bid, 12 weeks
  Arms: 2 Tranilast
Drug: Placebo — Placebo tablets, bid, 12 weeks
  Arms: 3

SUMMARY:
The purpose of this study is to evaluate whether tranilast at two different dosages compared to placebo is effective in patients with active RA when added to continuing methotrexate (MTX) therapy.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the efficacy and safety of two different doses of tranilast as determined by ACR20 response at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Receiving methotrexate
* Have at least 8 painful/tender and 6 swollen joints
* May be receiving oral steroids, chronic NSAIDs and/or hydroxychloroquine.

Exclusion Criteria:

* Use of any anti-arthritic treatments except those allowed in inclusion criteria
* Pregnant or nursing females
* Abnormal laboratory values
* History of clinically significant renal, hepatic dysfunction, psychiatric disorder, or alcohol/drug dependence
* Clinically significant systemic infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who achieve of ACR20 response | Week 12

SECONDARY OUTCOMES:
Proportion of subjects achieving ACR 50 and 70 response | Week 12
EULAR responders (e.g. DAS28 good or moderate responders) | week 12
Mean change from baseline of each ACR component | weeks 2, 4, 8, 12 and 16
Assess the safety and tolerability of both doses of tranilast | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kitt, MD, Study Director — Nuon Therapeutics, Inc.
Locations (32):
- United States (9):
  - Mesa, Arizona
  - Paradise Valley, Arizona
  - La Jolla, California
  - San Diego, California
  - Aventura, Florida
  - Frederick, Maryland
  - Lansing, Michigan
  - Hickory, North Carolina
  - Duncansville, Pennsylvania
- Argentina (4):
  - Capital Federal, Buenos Aires
  - Luján, Buenos Aires
  - Quilmes, Buenos Aires
  - Rosario, Santa Fe Province
- Bulgaria (2):
  - Plovdiv
  - Sofia
- Czechia (4):
  - Brno-Bohunice
  - Ostrava-Hlucin
  - Prague
  - Zlín
- Germany (6):
  - Hamburg
  - Ludwigsfelde
  - Naumburg
  - Osnabrück
  - Ratingen
  - Wiesbaden
- Mexico (4):
  - Mexicali, Estado de Baja California
  - Guadalajara, Jalisco
  - Morelia, Michoacán
  - Obregón, Sonora
- Serbia (2):
  - Belgrade
  - Niška Banja
- London, United Kingdom